CLINICAL TRIAL: NCT05252130
Title: Comparison of NoaScope to the Conventional Stethoscope for Auscultation of Heart and Lung Sounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innova Smart Technologies (Pvt.) Ltd (Other)
Collaborators: Rehman Medical Institute - RMI (Other); NOABIO LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NoaScope-1 RMI
Record Dates: First submitted 2021-12-24; First posted 2022-02-23 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Chest Pathology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Auscultation with a newly developed electronic stethoscope: NoaScope (Experimental): Identification of abnormal heart and lung sounds in study participants
  Interventions: Device: NoaScope

INTERVENTIONS:
Device: NoaScope — Smart digital stethoscope

SUMMARY:
Assessing non-inferiority of a newly developed electronic stethoscope NoaScope in comparison with the conventional 3M Littmann stethoscope

DETAILED DESCRIPTION:
The enrolled population will include adults with a history of heart and lung complications. The enhanced sound quality of the electronic stethoscope and its non-inferiority to the traditional/conventional 3M Littmann stethoscope will be assessed through auscultation examination of every patient by a health professional (consultant, medical resident, and house officer) with both the electronic stethoscope and 3M Littmann/traditional/conventional stethoscope

ELIGIBILITY:
Inclusion Criteria:

* Ages: 18 years or older (male and female)
* Hospital admitted or Out Patient Department
* Written consent provided

Exclusion Criteria:

* Age <18
* ICU admitted
* Written consent not provided

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Correctly identified abnormal heart and lung sounds by doctors using two stethoscopes: NoaScope and 3M™️ Littmann®️ Classic III. | 1 month
  Each patient will receive two auscultation examinations: one with NoaScope and another with 3M™️ Littmann®️ Classic III.
  The investigators will determine the clinical feasibility and non-inferiority of NoaScope to the FDA-approved 3M™️ Littmann®️ Classic III from auscultation findings (heart and lungs) by doctors (holding varied levels of clinical expertise). Doctors will examine each patient using two stethoscopes: NoaScope and 3M™️ Littmann®️ Classic III. The investigators will also measure inter and intra observer agreement by the Kappa index with the help of a questionnaire. Kappa values < 0.8 means weak to moderate level of agreement and Kappa values between 0.8 - 1.0 would mean strong level of agreement.
The measurement of sound quality in a clinical setting by means of an MOS scale on a questionnaire. | 1 month
  The investigators will measure sound quality on a mean opinion score scale with values ranging form 1 (bad) to 5 (excellent).

SECONDARY OUTCOMES:
Difference in performance between subgroups of doctors based on clinical experience. | 1 month
  This will be estimated as a proportion difference of correctly identified heart and lung sounds for each doctor subgroup.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehman Medical Institute - RMI, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No